CLINICAL TRIAL: NCT01863810
Title: Randomized, Double-blinded, Double-dummy, Active-controlled, Multi-center Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of KW21052 for 8 Weeks Compared to Pregabalin (Lyrica) in the Diabetic Patients With Neuropathic Pain
Brief Title: Efficacy and Safety of KW21052 Compared to Lyrica in the Diabetic Patients With Neuropathic Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KunWha Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KW21052_P3
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic Neuropathy; Neuropathic Pain; Pregabalin
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KW21052 (Experimental): This arm will be pre-treated with Lyrica 150mg (75mg bid) for titration period of 1 week and then be treated with KW21052 300mg and Placebo of Lyrica for intervention period of 8 weeks.
  Interventions: Drug: KW21052; Drug: Lyrica (low dose); Drug: Placebo of Lyrica
- LYRICA (Active Comparator): This arm will be pre-treated with Lyrica 150mg (75mg bid) for titration period of 1 week and then be treated with Lyrica 300mg (150mg bid) and Placebo of KW21052 300mg for intervention period of 8 weeks.
  Interventions: Drug: Lyrica; Drug: Lyrica (low dose); Drug: Placebo of KW21052

INTERVENTIONS:
Drug: KW21052 — 1 Tablet contains 300mg of pregabalin. Oral, once a day, for 8 weeks.
  Arms: KW21052
Drug: Lyrica — 1 Capsule contains 150mg of pregabalin. Oral, twice a day, for 8 weeks.
  Arms: LYRICA
Drug: Lyrica (low dose) — 1 Capsule contains 75mg of pregabalin. Oral, twice a day, for 1 week.
Drug: Placebo of KW21052 — Oral,once a day, for 8 weeks
  Arms: LYRICA
Drug: Placebo of Lyrica — Oral, twice a day, for 8 weeks.
  Arms: KW21052

SUMMARY:
Diabetic neuropathy is known to be the most common complication of diabetes, although the estimated prevalence is highly variable, ranging from 1.6 to 90%. Also, chronic pain is accompanied with sleep disorders, depression, and anxiety, thereby impairing quality of life and increasing societal costs. Pregabalin is one of proven and marketed oral medicine to manage the chronic neuropathic pain in diabetic patients. This study is designed as a randomized controlled trial to demonstrate that the efficacy of KW21052 in pain reduction measured by the weekly mean pain score on the numerical pain rating scale (NRS) at the 8th week of intervention is inferior to that of Lyrica.

DETAILED DESCRIPTION:
Patient Reported Outcomes (PRO) using validated questionnaires and patient diaries will be assessed for efficacy analysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and 2 diabetic patients
* Patients diagnosed with diabetic, distal, symmetrical, and sensorimotor polyneuropathy
* 40mm and more on VAS
* 4 and more on NRS
* Informed consented patients

Exclusion Criteria:

* Participating in another clinical trial
* Pregnancy or lactating
* Sensitivity to pregabalin
* Significant underlying disease or disorders
* Prohibited concomitant medications
* Significant laboratory abnormalities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale (NRS) | After 8 weeks of intervention

SECONDARY OUTCOMES:
Change on on the numerical pain rating scale (NRS) | From baseline to 8th week of intervention
Response rate | From baseline to 4th and 8th week of intervention
Clinical Global Impression of Change (CGIC) | After 8 weeks of intervention
Improved quality of life (QoL) | After 4 and 8 weeks of intervention
Drug compliance | During 8 weeks of intervention
Adverse events | Every clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Kuk Kim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea